CLINICAL TRIAL: NCT02901015
Title: Evaluation and Validation of Social Cognition Battery to Characterize Schizophrenic Patients Functioning (EVACO)
Brief Title: Evaluation and Validation of Social Cognition Battery to Characterize Schizophrenic Patients Functioning
Acronym: EVACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Eric BRUNET, Investigator coordinator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P11/34_EVACO
Record Dates: First submitted 2016-08-19; First posted 2016-09-15 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schizophrenic patients group 1 (Other): 80 patients evaluated in the Fondamental Expertise Center for schizophrenia Network (8 centers in France).
  Interventions: Behavioral: Assessment battery A
- Schizophrenic patients group 2 (Other): 80 patients evaluated in the Fondamental Expertise Center for schizophrenia Network (8 centers in France).
  Interventions: Behavioral: Assessment battery B

INTERVENTIONS:
Behavioral: Assessment battery A — Social cognition tests version "A" are administered to the patients
  Arms: Schizophrenic patients group 1
Behavioral: Assessment battery B — Social cognition tests version "B" are administered to the patients
  Arms: Schizophrenic patients group 2

SUMMARY:
Interventional, multicenter, and longitudinal study, of a cohort of patients with schizophrenia, evaluated on social cognition, neurocognition, symptoms, functioning with 12 months interval.

DETAILED DESCRIPTION:
The main objective is evaluation and validation of social cognition battery, characterizing the psychometric properties (validity, sensitivity to change) measures in a cohort of schizophrenic patients. Other objective is to demonstrate that the various components operating at T0 and T12 months of schizophrenic patients, as an external validator, are significantly explained by social cognition performance given the third known factors : neuropsychological, sociodemographic, disease course, and clinical status. Search and model relationships between the measured variables.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective disorder
* Age > 18 years and < 65 years
* Patient's state allows cognitive and neuropsychological assessment
* Affiliated to a social security system (beneficiary or legal).
* Informed consent signature (patients under guardianship may be included with written permission from their legal representative).

Exclusion Criteria:

* Alcohol dependence or current toxic
* Electroconvulsivotherapy (less than 6 months)
* Serious head trauma (become unconscious), epilepsy or neurological disorder significant or evolutionary
* Invalidating and uncorrected visual disorder
* Invalidating and not paired hearing
* Actually hospitalized under constraint
* Patient not able to come to different evaluations, or who plan to change medical care in the following year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in cognitive skills | Day 0, Month 12
  Change in the aggregates (average) of standardized performance levels : z-scores of Theory of mind (V-COMICS, V-SIR, SPEX), z-scores of empathy (QCAE), z-scores of facial affect recognition (TREF), z-scores of metacognition (V-COMICS meta), Intelligence quotient (WAIS-III), z-scores of treatment speed, z-scores of memory spans, z-scores of verbal memory, z-scores of visual memory, z-scores of attention/vigilance, z-scores of divided attention, z-scores of executive functions.

SECONDARY OUTCOMES:
Change in Functioning | Day 0, Month 12
  Change in the aggregates (average) of standardized functioning assessment: z-scores of social functioning, z-scores of general functioning (PSPS), and z-scores of help acceptance subscales (M-SEQ)
Change in Psychotic symptoms | Day 0, Month 12
  Change in the aggregates (average) of standardized symptomatology and clinical dimensions: z-scores of Schizophrenic syndromes, depressive syndrome and manic syndrome (PANSS), z-scores of observance scale (MARS/BARS), z-scores of insight (Birchwood), z-scores of antipsychotic medication doses

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - Hôpital Louis Mourier, Colombes
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Sainte Marguerite, Marseille
  - CHRU de Montpellier, Montpellier
  - Centre Hospitalier Alpes Isère, Saint Egrève
  - CHU de Strasbourg, Strasbourg